CLINICAL TRIAL: NCT04286867
Title: Examining Alcohol Consumption, Perceptions, and User Experience of Alcohol Moderation Strategies
Acronym: ALCMOD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kent State University (Other)
Responsible Party: Principal Investigator, William Lechner. PhD, Assistant Professor, Kent State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-199
Record Dates: First submitted 2020-02-21; First posted 2020-02-27 (Actual); Results first posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-09

CONDITIONS: Alcohol Abuse; Alcohol Use Disorder; Alcohol Abuse, Episodic
MeSH Terms: conditions — Alcoholism; Recurrence | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Two groups are defined and compared in terms of primary outcome measures.
Who Masked: Participant
Masking Description: All participants are told they will receive information about strategies and tools to reduce alcohol consumption. The participants will not be told whether they are receiving the novel method for reducing alcohol consumption or previously developed and studies methods for reducing alcohol consumption.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol Moderation Group 1 (Experimental): This group will receive a link and in-person instructions on how to use the alcohol moderation application described. This group will also receive training on the strategies for alcohol moderation recommended by NIAAA.
  Interventions: Other: Alcohol Moderation Mobile Application
- Alcohol Moderation Group 2 (Active Comparator): This group will receive the NIAAA tracking card and in-person instructions on how to use the drink tracker card (described at https://www.rethinkingdrinking.niaaa.nih.gov/Thinking-about-a-change/Strategies-for-cutting-down/Tips-To-Try.aspx). This group will also receive training on the strategies for alcohol moderation recommended by NIAAA.
  Interventions: Behavioral: Alcohol Moderation Drink Tracker

INTERVENTIONS:
Other: Alcohol Moderation Mobile Application — This group will receive a link and in-person instructions on how to use the alcohol moderation application described. Individuals in this group will define their drinking limits within the application. The application will provide time points to aid the individual in maintaining their predefined drinking limits throughout the course of the drinking occasion. This group will also receive training on the strategies for alcohol moderation recommended by NIAAA.
  Arms: Alcohol Moderation Group 1
Behavioral: Alcohol Moderation Drink Tracker — This group will receive the NIAAA tracking card and in-person instructions on how to use the drink tracker card (described at https://www.rethinkingdrinking.niaaa.nih.gov/Thinking-about-a-change/Strategies-for-cutting-down/Tips-To-Try.aspx). Individuals in this group will define their drinking limits, and record their alcohol consumption on the drink tracking card. This group will also receive training on the strategies for alcohol moderation recommended by NIAAA.
  Arms: Alcohol Moderation Group 2

SUMMARY:
The primary aims of the study are to assess the user experience and initial efficacy of a mobile application designed to reduce problematic alcohol use. The application utilizes drinking limits, defined by the user, to pace alcohol consumption during drinking occasions. The mobile application will be compared to strategies for tracking drinking detailed within the National Institute on Alcohol Abuse and Alcoholism Alcohol Moderation Strategies (https://www.rethinkingdrinking.niaaa.nih.gov/thinking-about-a-change/strategies-for-cutting-down/tips-to-try.aspx). Primary outcome variables, in addition to variables assessing user design experience of the application and use of moderation strategies, include (1) negative consequences of alcohol use during a 14 day observation period, and (2) number of drinks consumed per drinking day during a 14 day observation period.

DETAILED DESCRIPTION:
The mobile application to be tested provides guidance on moderating alcohol use in real time based on individual user's pre-defined drinking limits. This mobile application will be compared to a drink tracking strategy and corresponding tool outlined within the National Institute on Alcohol Abuse and Alcoholism Alcohol Moderation Strategies (https://www.rethinkingdrinking.niaaa.nih.gov/thinking-about-a-change/strategies-for-cutting-down/tips-to-try.aspx).

Participants will be recruited from the community in Northeastern Ohio. Eligible participants will meet the following inclusion criteria 1) be age 21 or older, 2) report experiencing at least three negative consequence of alcohol use in the past month (assessed via Brief Young Adult Alcohol Consequences Questionnaire: BYAACQ), 3) report having consumed at least 5 drinks (for men) or 4 drinks (for women) on one or more occasions in the past 2-weeks, 4) not be seeking treatment for alcohol use from a health-care provider, and 5) have access to a smartphone and 6) endorse some importance in changing their drinking (2 or greater on Alcohol Ladder Scale Importance to Change). Participants who endorse seeking treatment for alcohol related problems from a health care provider will be provided with a list of university sponsored and community based treatment providers, and excluded. Participants (n=64) will complete a battery of assessments including demographic measures, alcohol and substance use measures, psychological measures, behavioral economic and neuropsychological measures.

The Timeline Follow-back Interview will be used to assess alcohol use. The Brief Young Adult Alcohol Consequences Questionnaire (BYAACQ ) will be used to assess a range of negative consequences of alcohol use that young adults may experience (e.g., while drinking in the past month, I have said or done embarrassing things).

Following this initial baseline assessment, participants will be randomized to one of two experimental conditions detailed below (Alcohol Moderation Group 1 and 2). Doctoral Candidates in Clinical Psychology will review strategies for moderating alcohol use with all participants (strategies recommended by the National Institute on Alcohol Abuse and Alcoholism; detail included as supplement). The only variation in the discussion of strategies is the the Alcohol Moderation Group 1 will receive detail and training on how to use the mobile application; whereas, the Alcohol Moderation Group 2 will receive detail and training on how to use the drinking tracker card recommended within the NIAAA guidelines.

Primary outcome variables, in addition to variables assessing user design experience of the application and use of moderation strategies, will include (1) negative consequences of alcohol use during a 14 day observation period following randomization, and (2) number of drinks consumed per drinking day during a 14 day observation period following randomization. Assessment of primary outcome variable (1) will include baseline negative consequences of alcohol use (BYAACQ score) during the 14 day period prior to randomization as a covariate as well as additional covariates defined a priori based on the extant literature. Assessment of primary outcome variable (2) will include consideration of average drinking limit for each drinking day defined by the user, and number of drinks per drinking day in a 14 day period prior to randomization, as well as covariates defined a priori based on the extant literature.

ELIGIBILITY:
Inclusion Criteria:

1. must report experiencing at least three negative consequences of alcohol use in the past month (assessed via Brief Young Adult Alcohol Consequences Questionnaire: BYAACQ)
2. have access to a smartphone
3. endorse importance in changing their drinking (2 or greater on Alcohol Ladder Scale Importance to Change)
4. report having consumed at least 5 drinks (for men) or 4 drinks (for women) on one or more occasions in the past 2-weeks

Exclusion Criteria:

1. seeking treatment for alcohol use from a health-care provider
2. younger than age 21

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kent State University, Kent, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alcohol Moderation Group 1 | Alcohol Moderation Group 2
Started | 32 | 32
Completed | 29 | 30
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcohol Moderation Group 1 | Alcohol Moderation Group 2 | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.11 (16.05) | 38.41 (14.25) | 37.77 (15.05)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Identified Gender: Female | 23 | 21 | 44
  Identified Gender: Male | 5 | 9 | 14
  Identified Gender: Identified as another gender | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 28 | 28 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 27 | 27 | 54
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 29 | 30 | 59

OUTCOME MEASURES:

1. Primary Outcome: The Young Adult Alcohol Consequences Questionnaire
Description: The Brief Young Adult Alcohol Consequences Questionnaire (BYAACQ) will be used to assess negative consequences of alcohol use (24-items). Minimum score is 0, maximum is 24, with higher scores indicating more negative consequences of alcohol use.
Time Frame: 14 day window preceding baseline assessed at baseline, 14 day window assessed 14 days following baseline
Measure: Mean (Standard Deviation); unit: outcome score minus baseline score
Arm/Group | Alcohol Moderation Group 1 | Alcohol Moderation Group 2
Number analyzed (Participants) | 29 | 30
outcome score minus baseline score | -4.48 (4.07) | -4.63 (3.97)

2. Primary Outcome: Number of Standard Drinks Consumed Per Drinking Day
Description: A daily alcohol use diary will be provided for the two-week observation period. Participants will be trained on how to use the diary during the baseline laboratory session. Number of standard drinks per drinking day will be calculated from the daily diary alcohol consumption records (total number of standard drinks consumed / number of drinking days).
Time Frame: 14 day window preceding baseline assessed at baseline, 14 day window assessed 14 days following baseline
Measure: Mean (Standard Deviation); unit: change in standard drinks
Arm/Group | Alcohol Moderation Group 1 | Alcohol Moderation Group 2
Number analyzed (Participants) | 28 | 30
change in standard drinks | -.618 (1.81) | -.955 (2.21)

ADVERSE EVENTS:
Time Frame: each participant was assessed for adverse events from the time of their consent to intitate the study until the end of the final outcome session in which assessments were collected, 14 days in total.
Arm/Group | Alcohol Moderation Group 1 | Alcohol Moderation Group 2
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/29 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-05-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT04286867/Prot_ICF_000.pdf